CLINICAL TRIAL: NCT03444402
Title: A Randomized, Open-label, Multiple-dose, and Three-way Crossover Clinical Trial to Compare Pharmacokinetics and Safety of CKD-381 and D026 in Healthy Male Subjects
Brief Title: A Study to Compare PK and Safety of CKD-381 and D026 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 173HPS17013
Record Dates: First submitted 2018-02-06; First posted 2018-02-23 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: GERD
Keywords: CKD-381; Nexium
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Period 1: Test drug(CKD-381 formulation I), Period 2: Test drug(CKD-381 formulation II), Period 3: Reference drug(D026)
  Interventions: Drug: CKD-381(formulation I); Drug: CKD-381(formulation II); Drug: D026(Nexium 40mg)
- Group B (Experimental): Period 1: Test drug(CKD-381 formulation II), Period 2: Reference drug(D026), Period 3: Test drug(CKD-381 formulation I)
  Interventions: Drug: CKD-381(formulation I); Drug: CKD-381(formulation II); Drug: D026(Nexium 40mg)
- Group C (Experimental): Period 1: Reference drug(D026), Period 2: Test drug(CKD-381 formulation I), Period 3: Test drug(CKD-381 formulation II)
  Interventions: Drug: CKD-381(formulation I); Drug: CKD-381(formulation II); Drug: D026(Nexium 40mg)

INTERVENTIONS:
Drug: CKD-381(formulation I) — 1 tablet administered before the breakfast during 7 days
Drug: CKD-381(formulation II) — 1 tablet administered before the breakfast during 7 days
Drug: D026(Nexium 40mg) — 1 tablet administered before the breakfast during 7 days

SUMMARY:
A Study to compare pharmacokinetics and safety of CKD-381 and D026 in healthy male subjects

DETAILED DESCRIPTION:
A randomized, open-label, multiple-dose, and three-way cross over clinical trial to compare pharmacokinetics and safety of CKD-381 and D026 in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 aged and 50 aged in healthy male adult
2. Body weight more than 55kg
3. Body Mass Index more than 18.5 and under 25

Exclusion Criteria:

1. Have clinically significant disease that hepatobiliary system, kidney, nervous system, immune system, respiratory system, endocrine system, hemato-oncology disease, cardiovascular system or mental illness, or a history of mental disease.
2. Have a gastrointestinal disease history that can effect drug absorption or surgery.
3. Hypersensitivity reaction or clinically significant hypersensitivity reaction in the history of Esomeprazole, additives or benzimidazole family.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
AUCtau,ss(Area under the plasma drug concentration-time curve within a dosing interval at steady state) | 0~24h
  Evaluation PK esomeprazole after multiple dose

SECONDARY OUTCOMES:
Cmax,ss(Maximum concentration of drug in plasma at steady state) | 0~24h
  Evaluation PK esomeprazole after multiple dose
Tmax,ss(Time to maximum plasma concentration at steady state) | 0~24h
  Evaluation PK esomeprazole after multiple dose
t1/2(Terminal elimination half-life) | 0~24h
  Evaluation PK esomeprazole after multiple dose
R(Accumulation ratio) | 0~24h
  Evaluation PK esomeprazole after multiple dose
CLss/F(Apparent Clearance at steady state) | 0~24h
  Evaluation PK esomeprazole after multiple dose
Vss/F(Apparent Volume of distribution at steady state) | 0~24h
  Evaluation PK esomeprazole after multiple dose
Cmax(Maximum concentration of drug in plasma) | 0~24h
  Evaluation PK esomeprazole after single dose
AUClast(Area under the plasma drug concentration-time curve from 0 to last) | 0~24h
  Evaluation PK esomeprazole after single dose
Tmax(Time to maximum plasma concentration) | 0~24h
  Evaluation PK esomeprazole after single dose
t1/2(Terminal elimination half-life) | 0~24h
  Evaluation PK esomeprazole after single dose
CL/F(Apparent clearance) | 0~24h
  Evaluation PK esomeprazole after single dose
Vd/F(Apparent volume of distribution) | 0~24h
  Evaluation PK esomeprazole after single dose

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Sang Yu, M.D, Principal Investigator — Department of Clinical Pharmacology and Therapeutics, Seoul National University College of Medicine and Hospital
Locations (1):
- Seoul University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No